CLINICAL TRIAL: NCT02346994
Title: Development and Expansion of Melt Organic Baking Fat for Oxidative Stability and Reducing Child Obesity
Brief Title: Development of Melt Organic Baking Fat for Reducing Child Obesity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: United States Department of Agriculture (USDA) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Marie-Pierre St-Onge, Assistant Professor, Columbia University
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AAAN3253; NCT02132377 (obsolete NCT alias)
Record Dates: First submitted 2015-01-16; First posted 2015-01-27 (Estimated); Last update posted 2017-01-31 (Estimated); Status verified 2017-01

CONDITIONS: Obesity; Overweight; Pediatric Obesity
Keywords: Body Weight; Obesity in Adolescence; Obesity in Childhood; Childhood Onset Obesity; Childhood Obesity; Child Obesity; Adolescent Obesity; Teenagers; Teens; Youth; Adolescents; Adolescence
MeSH Terms: conditions — Obesity; Overweight; Pediatric Obesity; Body Weight | interventions — Corn Oil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Melt test blend 3.2 (Experimental)
  Interventions: Dietary Supplement: Melt Test Blend 3.2
- Corn Oil (Active Comparator)
  Interventions: Dietary Supplement: Corn Oil

INTERVENTIONS:
Dietary Supplement: Melt Test Blend 3.2 — Participant will be given a standard breakfast (containing 20 g of fat from test blend 3.2) to consume over a 10-min period. Test blend 3.2 will be provided in test muffins. The test breakfast will provide 35% of the participant's daily energy requirements, estimated using the Schofield equation. The muffin will provide 450 kcal, and the rest of the energy will be in the form of fat free yogurt, up to 140 kcal, and applesauce.
  Arms: Melt test blend 3.2
Dietary Supplement: Corn Oil — Participant will be given a standard breakfast (containing 20 g of fat from corn oil) to consume over a 10-min period. Corn oil will be provided in test muffins. The test breakfast will provide 35% of the participant's daily energy requirements, estimated using the Schofield equation. The muffin will provide 450 kcal, and the rest of the energy will be in the form of fat free yogurt, up to 140 kcal, and applesauce.
  Arms: Corn Oil

SUMMARY:
The purpose of this study is to compare the effects of a cooking oil on metabolic rate, appetite, and metabolic risk markers.

DETAILED DESCRIPTION:
The overall objectives of this study are to determine whether a Melt Organic baking blend can alter energy balance towards a negative energy balance by enhancing thermic effect of food and improving feelings of satiety relative to a control, corn oil, in overweight and obese adolescents.

This study will employ a 2-arm, double-blind, randomized, crossover design. Each arm will consist of one test day and will differ in the type of oil incorporated in the test breakfast: test blend 3.2 or corn oil. Oil sequence will be randomized. Each test day will follow the same protocol and will be separated by at least two weeks for boys or 4 weeks for girls to ensure that testing occurs during the same phase of their menstrual cycle for each test day.

Participants will arrive at the testing center after an overnight 12-h fast. Upon arrival, body weight will be taken and a catheter will be inserted in an antecubital vein. The participant will then rest for 30 minutes, after which resting metabolic rate (RMR) will be measured using an indirect calorimetry cart. RMR will be measured over a 45-min period. At the end of the RMR measurement, a fasting blood sample will be obtained, and the participant will be given a standard breakfast (containing 20 g of fat from either test blend 3.2 or corn oil) to consume over a 10-min period. The fat in the breakfast will be provided in test muffins. The test breakfast will provide 35% of the participant's daily energy requirements, estimated using the Schofield equation. The muffin will provide 450 kcal and the rest of the energy will be provided in the form of fat free yogurt, up to 140 kcal, and applesauce.

Following breakfast, postprandial energy expenditure will be assessed every hour using the indirect calorimetry cart. At each hour of this 5-h period, participants will fill out a visual analog scale to assess their feelings of appetite and satiety and will perform a computer task assessing prospective food intake. Immediately after breakfast, and at 30, 45, 60, 120, and 180 minutes after breakfast, a blood sample will be drawn from the catheter for metabolite and hormone measurements.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index (BMI) equal to or greater than 85th percentile for age and sex
* Weight stable (+/- 2.5 kg) for at least 3 months prior to screening

Exclusion Criteria:

* Any endocrine disorder, including type 1 diabetes
* Weight loss attempted in past 3 months
* Currently using medication (prescription or over-the-counter) that could impact study outcomes
* Asthma
* Anemia
* Diagnosis of psychoses, bipolar disorder, major depression, severe personality disorder; history of suicidal tendencies
* Use of (current or in the past 4 weeks) any investigational medications or devices
* Allergy/sensitivity to wheat, milk, eggs, nuts

Ages: 15 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 15 (Actual)
Dates: Start 2013-01; Primary Completion 2016-08 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Thermic effect of food | 5.5 hours
  An indirect calorimetry cart will measure energy expenditure for approximately 40 minutes out of each hour for 5 hours after breakfast.

SECONDARY OUTCOMES:
Appetite/satiety measures area under the curve | 5.5 hours
  A visual analog scale and a computer program will assess different aspects of appetite and satiety in study participants.
Insulin, glucose, triglycerides area under the curve | Fasting, and at minutes 0, 30, 45, 60, 120, and 180 after the end of breakfast
  Blood draw and analyses will be used to measure triglycerides, glucose, and insulin.

CONTACTS AND LOCATIONS:
Overall Officials: Marie-Pierre St-Onge, Ph.D., Principal Investigator — Columbia University
Locations (1):
- New York Nutrition Obesity Research Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided